CLINICAL TRIAL: NCT03998332
Title: Overall Survival and Progression Free Survival of Patients With Large Cell Neuroendocrine Lung Cancer and Combined Large Cell Neuroendocrine Lung Cancer Treated in Clinical Stage I-IV
Brief Title: Overall Survival of Large Cell Neuroendocrine Lung Cancer Patients - a Retrospective Study
Status: Completed | Type: Observational
Sponsor: Jaroslaw B. Cwikla, MD, PhD, Professor UWM (Other)
Responsible Party: Sponsor-Investigator, Jaroslaw B. Cwikla, MD, PhD, Professor UWM, Head of Department of Radiology, University of Warmia and Mazury
Organization: University of Warmia and Mazury (Other)
Other Study IDs: LCNEC_2018
Record Dates: First submitted 2019-06-18; First posted 2019-06-26 (Actual); Last update posted 2019-07-01 (Actual); Status verified 2019-06

CONDITIONS: Survival Outcomes of Patients With Pulmonary LCNEC
Keywords: LCNEC-Large cell neuroendocrine carcinoma; Lung cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a retrospective study. 132 patients with LCNEC and combined LCNEC were included to the analysis. Patients were treated with radical, palliative or symptomatic intension between 2002-2018 in central and north-eastern centres in Poland. The group of patients consists of 47 women (36%) and 85 men (64%). Ratio of women to men is 1:1,81. The observation period ranged from 0 to 192 months.

DETAILED DESCRIPTION:
This is a retrospective study. 132 patients with LCNEC and combined LCNEC were included to the analysis. Patients were treated with radical, palliative or symptomatic intension between 2002-2018 in central and north-eastern centres in Poland. The group of patients consists of 47 women (36%) and 85 men (64%). Ratio of women to men is 1:1,81. The observation period ranged from 0 to 192 months.

For all patients included to the analysis, the clinical stage was estimated according to TNM Classification of Malignant Tumours - UICC from 2017. The degree of pathomorphic stage (pTNM) was assessed in 60 patients treated with intention to treat (ITT), which is 45% of the total population.

The degree of clinical stage (cTNM) was assessed in 72 patients based on the imaging examinations (including PET, CT, MRI, bone scintigraphy, etc.) and fine needle aspiration biopsy (FNA) (including EBUS, with pathological confirmation of LCNEC, which is 55% of the total population.

The clinical stage (cTNM) was used in case of patients disqualified from radical surgery due to: advanced disease, contraindications to surgery, no patient's consent for treatment.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥18 years old, male or female, with pathologically confirmed primary neuroendocrine lung cancer based on histopathological examination:

  1. LCNEC
  2. combined type LCNEC
* Patients with LCNEC, combined LCNEC without prior treatment independently from the clinical stage according to the 8th edition of TNM 2017
* Patients with generalized, unresectable of LCNEC, combined LCNEC before, during and after palliative treatment
* Patients with generalized, unresectable LCNEC, combined LCNEC treated only symptomatically
* Patients with locally advanced, unresectable LCNEC,combined LCNEC before, during and after radical treatment
* Patients with locally advanced, resectable LCNEC, combined LCNEC before, during and after treatment

Exclusion Criteria:

* NA

Ages: 18 Years to 86 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 132 patients with LCNEC and combined LCNEC were included to the analysis. Patients were treated with radical, palliative or symptomatic intension between 2002-2018 in central and north-eastern centres in Poland. The group of patients consists of 47 women (36%) and 85 men (64%). Ratio of women to men is 1:1,81. The observation period ranged from 0 to 192 months.
Sampling Method: Non-Probability Sample
Enrollment: 132 (Actual)
Dates: Start 2002-01-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
PFS - Progression Free Survival | 16 years
  the time from the start of treatment date to the date of first observation of documented local recurrence, metastases or disease progression. Patients without progression at the time of analysis will be censored.
OS - Overall Survival | 16 years
  is defined as the time from the histopathological confirmation to the date of death due to any cause or the date of last contact (censored observation) at the date of data cut-off.

SECONDARY OUTCOMES:
Log-rank test | 16 years
  assessment of differences in survival of patients between subgroups
Cox proportional-hazards model | 16 years
  multivariate analyses used for investigating the association between the survival time of patients and prognostic factors

CONTACTS AND LOCATIONS:
Overall Officials: Jarosław B Ćwikła, MD, PhD, Study Chair — University of Warmia and Mazury

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Rekhtman N. Neuroendocrine tumors of the lung: an update. Arch Pathol Lab Med. 2010 Nov;134(11):1628-38. doi: 10.5858/2009-0583-RAR.1. PMID 21043816
- [Result] Travis WD. Advances in neuroendocrine lung tumors. Ann Oncol. 2010 Oct;21 Suppl 7:vii65-71. doi: 10.1093/annonc/mdq380. PMID 20943645
- [Result] Gustafsson BI, Kidd M, Chan A, Malfertheiner MV, Modlin IM. Bronchopulmonary neuroendocrine tumors. Cancer. 2008 Jul 1;113(1):5-21. doi: 10.1002/cncr.23542. PMID 18473355
- [Result] Detterbeck FC. Management of carcinoid tumors. Ann Thorac Surg. 2010 Mar;89(3):998-1005. doi: 10.1016/j.athoracsur.2009.07.097. PMID 20172187
- [Result] Wolin EM. Challenges in the Diagnosis and Management of Well-Differentiated Neuroendocrine Tumors of the Lung (Typical and Atypical Carcinoid): Current Status and Future Considerations. Oncologist. 2015 Oct;20(10):1123-31. doi: 10.1634/theoncologist.2015-0198. Epub 2015 Aug 25. PMID 26306904
- [Result] Chong CR, Wirth LJ, Nishino M, Chen AB, Sholl LM, Kulke MH, McNamee CJ, Janne PA, Johnson BE. Chemotherapy for locally advanced and metastatic pulmonary carcinoid tumors. Lung Cancer. 2014 Nov;86(2):241-6. doi: 10.1016/j.lungcan.2014.08.012. Epub 2014 Aug 27. PMID 25218177
- [Result] Modlin IM, Oberg K, Chung DC, Jensen RT, de Herder WW, Thakker RV, Caplin M, Delle Fave G, Kaltsas GA, Krenning EP, Moss SF, Nilsson O, Rindi G, Salazar R, Ruszniewski P, Sundin A. Gastroenteropancreatic neuroendocrine tumours. Lancet Oncol. 2008 Jan;9(1):61-72. doi: 10.1016/S1470-2045(07)70410-2. PMID 18177818
- [Result] Modlin IM, Lye KD, Kidd M. A 5-decade analysis of 13,715 carcinoid tumors. Cancer. 2003 Feb 15;97(4):934-59. doi: 10.1002/cncr.11105. PMID 12569593
- [Result] Yao JC, Hassan M, Phan A, Dagohoy C, Leary C, Mares JE, Abdalla EK, Fleming JB, Vauthey JN, Rashid A, Evans DB. One hundred years after "carcinoid": epidemiology of and prognostic factors for neuroendocrine tumors in 35,825 cases in the United States. J Clin Oncol. 2008 Jun 20;26(18):3063-72. doi: 10.1200/JCO.2007.15.4377. PMID 18565894
- [Result] Vinik AI, Woltering EA, Warner RR, Caplin M, O'Dorisio TM, Wiseman GA, Coppola D, Go VL; North American Neuroendocrine Tumor Society (NANETS). NANETS consensus guidelines for the diagnosis of neuroendocrine tumor. Pancreas. 2010 Aug;39(6):713-34. doi: 10.1097/MPA.0b013e3181ebaffd. No abstract available. PMID 20664471
- [Result] Oberg K, Hellman P, Ferolla P, Papotti M; ESMO Guidelines Working Group. Neuroendocrine bronchial and thymic tumors: ESMO Clinical Practice Guidelines for diagnosis, treatment and follow-up. Ann Oncol. 2012 Oct;23 Suppl 7:vii120-3. doi: 10.1093/annonc/mds267. No abstract available. PMID 22997444
- [Result] Caplin ME, Baudin E, Ferolla P, Filosso P, Garcia-Yuste M, Lim E, Oberg K, Pelosi G, Perren A, Rossi RE, Travis WD; ENETS consensus conference participants. Pulmonary neuroendocrine (carcinoid) tumors: European Neuroendocrine Tumor Society expert consensus and recommendations for best practice for typical and atypical pulmonary carcinoids. Ann Oncol. 2015 Aug;26(8):1604-20. doi: 10.1093/annonc/mdv041. Epub 2015 Feb 2. PMID 25646366
- [Result] Fisseler-Eckhoff A, Demes M. Neuroendocrine tumors of the lung. Cancers (Basel). 2012 Jul 31;4(3):777-98. doi: 10.3390/cancers4030777. PMID 24213466
- [Result] Detterbeck FC. Clinical presentation and evaluation of neuroendocrine tumors of the lung. Thorac Surg Clin. 2014 Aug;24(3):267-76. doi: 10.1016/j.thorsurg.2014.04.002. PMID 25065927
- [Result] Pieterman CR, Conemans EB, Dreijerink KM, de Laat JM, Timmers HT, Vriens MR, Valk GD. Thoracic and duodenopancreatic neuroendocrine tumors in multiple endocrine neoplasia type 1: natural history and function of menin in tumorigenesis. Endocr Relat Cancer. 2014 May 6;21(3):R121-42. doi: 10.1530/ERC-13-0482. Print 2014 Jun. PMID 24389729
- [Result] Aguayo SM, Miller YE, Waldron JA Jr, Bogin RM, Sunday ME, Staton GW Jr, Beam WR, King TE Jr. Brief report: idiopathic diffuse hyperplasia of pulmonary neuroendocrine cells and airways disease. N Engl J Med. 1992 Oct 29;327(18):1285-8. doi: 10.1056/NEJM199210293271806. No abstract available. PMID 1406819
- [Result] Gosney JR. Diffuse idiopathic pulmonary neuroendocrine cell hyperplasia as a precursor to pulmonary neuroendocrine tumors. Chest. 2004 May;125(5 Suppl):108S. doi: 10.1378/chest.125.5_suppl.108s. No abstract available. PMID 15136447
- [Result] Koo CW, Baliff JP, Torigian DA, Litzky LA, Gefter WB, Akers SR. Spectrum of pulmonary neuroendocrine cell proliferation: diffuse idiopathic pulmonary neuroendocrine cell hyperplasia, tumorlet, and carcinoids. AJR Am J Roentgenol. 2010 Sep;195(3):661-8. doi: 10.2214/AJR.09.3811. PMID 20729444
- [Result] Chong S, Lee KS, Chung MJ, Han J, Kwon OJ, Kim TS. Neuroendocrine tumors of the lung: clinical, pathologic, and imaging findings. Radiographics. 2006 Jan-Feb;26(1):41-57; discussion 57-8. doi: 10.1148/rg.261055057. PMID 16418242
- [Result] Travis WD, Rush W, Flieder DB, Falk R, Fleming MV, Gal AA, Koss MN. Survival analysis of 200 pulmonary neuroendocrine tumors with clarification of criteria for atypical carcinoid and its separation from typical carcinoid. Am J Surg Pathol. 1998 Aug;22(8):934-44. doi: 10.1097/00000478-199808000-00003. PMID 9706973
- [Result] Igawa S, Watanabe R, Ito I, Murakami H, Takahashi T, Nakamura Y, Tsuya A, Kaira K, Naito T, Endo M, Yamamoto N, Kameya T. Comparison of chemotherapy for unresectable pulmonary high-grade non-small cell neuroendocrine carcinoma and small-cell lung cancer. Lung Cancer. 2010 Jun;68(3):438-45. doi: 10.1016/j.lungcan.2009.07.003. Epub 2009 Aug 21. PMID 19699548
- [Result] Watanabe R, Ito I, Kenmotsu H, Endo M, Yamamoto N, Ohde Y, Kondo H, Nakajima T, Kameya T. Large cell neuroendocrine carcinoma of the lung: is it possible to diagnose from biopsy specimens? Jpn J Clin Oncol. 2013 Mar;43(3):294-304. doi: 10.1093/jjco/hys221. Epub 2013 Feb 3. PMID 23381206
- [Result] Kujtan L, Muthukumar V, Kennedy KF, Davis JR, Masood A, Subramanian J. The Role of Systemic Therapy in the Management of Stage I Large Cell Neuroendocrine Carcinoma of the Lung. J Thorac Oncol. 2018 May;13(5):707-714. doi: 10.1016/j.jtho.2018.01.019. Epub 2018 Jan 31. PMID 29391287
- [Result] Hiroshima K, Mino-Kenudson M. Update on large cell neuroendocrine carcinoma. Transl Lung Cancer Res. 2017 Oct;6(5):530-539. doi: 10.21037/tlcr.2017.06.12. PMID 29114469
- [Result] Yang G, Pan Z, Ma N, Qu L, Yuan T, Pang X, Yang X, Dong L, Liu S. Leptomeningeal metastasis of pulmonary large-cell neuroendocrine carcinoma: A case report and review of the literature. Oncol Lett. 2017 Oct;14(4):4282-4286. doi: 10.3892/ol.2017.6676. Epub 2017 Jul 26. PMID 28943940
- [Result] Ramirez RA, Chauhan A, Gimenez J, Thomas KEH, Kokodis I, Voros BA. Management of pulmonary neuroendocrine tumors. Rev Endocr Metab Disord. 2017 Dec;18(4):433-442. doi: 10.1007/s11154-017-9429-9. PMID 28868578
- [Result] Tang H, Wang H, Xi S, He C, Chang Y, Wang Q, Wu Y. Perioperative chemotherapy with pemetrexed and cisplatin for pulmonary large-cell neuroendocrine carcinoma: a case report and literature review. Onco Targets Ther. 2018 May 7;11:2557-2563. doi: 10.2147/OTT.S160565. eCollection 2018. PMID 29765234
- [Result] Derks JL, van Suylen RJ, Thunnissen E, den Bakker MA, Groen HJ, Smit EF, Damhuis RA, van den Broek EC, Speel EM, Dingemans AC; PALGA group. Chemotherapy for pulmonary large cell neuroendocrine carcinomas: does the regimen matter? Eur Respir J. 2017 Jun 1;49(6):1601838. doi: 10.1183/13993003.01838-2016. Print 2017 Jun. PMID 28572122
- [Result] Prelaj A, Rebuzzi SE, Del Bene G, Giron Berrios JR, Emiliani A, De Filippis L, Prete AA, Pecorari S, Manna G, Ferrara C, Rossini D, Longo F. Evaluation of the efficacy of cisplatin-etoposide and the role of thoracic radiotherapy and prophylactic cranial irradiation in LCNEC. ERJ Open Res. 2017 Mar 29;3(1):00128-2016. doi: 10.1183/23120541.00128-2016. eCollection 2017 Jan. PMID 28382303
- [Result] Kim KW, Kim HK, Kim J, Shim YM, Ahn MJ, Choi YL. Outcomes of Curative-Intent Surgery and Adjuvant Treatment for Pulmonary Large Cell Neuroendocrine Carcinoma. World J Surg. 2017 Jul;41(7):1820-1827. doi: 10.1007/s00268-017-3908-8. PMID 28204910